CLINICAL TRIAL: NCT04984070
Title: Research on Risk Factors and Comprehensive Intervention Measures of Polycystic Ovary Syndrome Complicated With Mental Diseases Such as Depression and Anxiety
Brief Title: Research on Risk Factors and Interventions of Polycystic Ovary Syndrome Complicated With Depression and Anxiety
Acronym: PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhang Wei, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FudanU2021-07-19
Record Dates: First submitted 2021-07-24; First posted 2021-07-30 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Depression, Anxiety
Keywords: polycystic ovary syndrome; depression; anxiety; bipolar disorder; intervention
MeSH Terms: conditions — Polycystic Ovary Syndrome; Depression; Anxiety Disorders; Bipolar Disorder | interventions — Contraceptives, Oral, Combined; drospirenone; Ethinyl Estradiol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCOS treatment (Experimental): Lifestyle intervention, oral contraceptive pills and metformin will be given to improve the symptoms of PCOS patients, such as obesity, hyperandrogegism, and insulin resistance, and to compare the different psychological status in PCOS.
  Interventions: Drug: Oral Contraceptives, Combined; Drug: Metformin Pill; Other: lifestyle intervention

INTERVENTIONS:
Drug: Oral Contraceptives, Combined — One of the three medications like ethinylestradiol (35 μg) and cyproterone acetate, drospirenone and ethinylestradiol tablets (I) and (Ⅱ) will be used as an antiandrogen.
  Other Names: Danie-35; Drospirenone and Ethinylestradiol Tablets (I); Drospirenone and Ethinylestradiol Tablets (Ⅱ)
Drug: Metformin Pill — Metformin is used to lower insulin resistance or to modulate hyperinsulinism.
  Other Names: Metformin
Other: lifestyle intervention — Weight control including calorie restriction and moderate exercise will be recommended to obese PCOS patients

SUMMARY:
The current study intends to establish a prediction method and evaluation system for polycystic ovary syndrome (PCOS) complicated with affective disorder, such as depression and anxiety, through the epidemiological investigation. Randomized controlled studies on the efficacy of various intervention methods should be carried out to develop early intervention measures and methods in order to reduce the harm of psychological disorders, to facilitate the mental health of PCOS patients, and thus to improve the quality of life.

DETAILED DESCRIPTION:
PCOS is one of the most common reproductive endocrine and metabolic diseases in women of adolescence and childbearing age. The prevalence of PCOS in reproductive women is as high as 5-10%, about 50-80% of whom are infertile and need ovulation induction or in vitro fertilization-embryo transfer (IVF-ET). Ovulation/anovulation and hyperandrogenemia are two main features of PCOS. Moreover, about 50-60% of PCOS patients present insulin resistance/hyperinsulinemia. The probability of miscarriage in PCOS is also higher than that of control women. Pregnancy complications in PCOS patients, such as gestational diabetes, preeclampsia, etc., and long-term complications of metabolic syndrome and endometrial cancer are more likely to happen. These not only greatly affect women's reproductive health, but also seriously endanger their psychological status. A large sample of data has shown that the risk of depression in women with PCOS is 3.78 times higher than that of the control women, 5.62 times for anxiety, and 1.78 times for bipolar disorder. With the economic development, more and more attention is paid to the quality of life including their mental health. However, there is few data on the risk factors of depression, anxiety and other psychological disorders in women with PCOS. There is a lack of effective evaluation and prediction systems. It is urgent to establish a risk assessment system for PCOS complicated with psychological diseases through scientific and systematic research, to formulate comprehensive intervention measures to improve the quality of life of women with PCOS and to reduce the incidence of affective disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as PCOS according to Rotterdam criteria 2003, aged between 18 and 40 years old, and no willing to get pregnant in a year.

At least two of the following three criteria were met: clinical and/or biochemical signs of hyperandrogenism, oligo- and/or anovulation, and polycystic ovary on ultrasonography,

Exclusion Criteria:

* Any other related diseases, such as adrenal congenital hyperplasia, Cushing's syndrome, androgen-secreting tumors, Hashimoto's thyroiditis, hyperthyroidism or hypothyroidism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | one year
  The self-rating depression scale(SDS) is assessed before and after intervention. The SDS score multiplied by 1.25 is a standard score, which is between 25-100. A score no less than 50 is consider as depression.
Anxiety | one year
  The self-rating anxiety scale(SAS) is assessed before and after intervention. The SAS score multiplied by 1.25 is a standard score, which is between 25-100. A score no less than 50 is consider as anxiety.
Health Related Quality of Life in PCOS | one year
  The scores of Health Related Quality of Life Questionnaire are assessed before and after treatment, which range from 30 to 210. Higher scores indicate higher quality of life of PCOS patients with less influence from PCOS.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Doctor, Study Director — OB & GYN Hospital of Fudan University
Locations (1):
- OB & GYN Hospital of Fudan University, Shanghai, Shanghai Municipality, China